CLINICAL TRIAL: NCT03829007
Title: PINCH - PD-L1 ImagiNg to prediCt Durvalumab Treatment Response in HNSCC
Brief Title: PD-L1 ImagiNg to prediCt Durvalumab Treatment Response in HNSCC
Acronym: PINCH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PINCH
Record Dates: First submitted 2019-01-09; First posted 2019-02-04 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Head and Neck Cancer
Keywords: durvalumab; PD-L1 imaging
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 imaging (Experimental): 89Zr-durvalumab iv injection followed by a PET/CT scan at day 5 after injection.
  Interventions: Diagnostic Test: PD-L1 imaging; Drug: Durvalumab

INTERVENTIONS:
Diagnostic Test: PD-L1 imaging — 89Zr-durvalumab injection followed by a PET/CT scan 5 days after injection
  Other Names: 89Zr-durvalumab PET/CT
Drug: Durvalumab — Durvalumab treatment is initiated after the PET/CT scan in a fixed dose of 1500 mg iv q4w

SUMMARY:
Non-invasive imaging of tumor PD-L1 expression with 89Zr-labeled durvalumab PET/CT predicts response to durvalumab.

DETAILED DESCRIPTION:
The programmed death 1 (PD1)/ programmed death ligand 1 (PD-L1) pathway plays an important role in regulating the T-cell anti tumor response. Blocking this interaction with the anti PD-L1 monoclonal antibody durvalumab has proven to be effective resulting in durable disease control rates. Currently, PD-L1 expression as determined by immune histochemistry (IH) is the best available biomarker for treatment response, but standardized scoring criteria are lacking and the risk for sampling errors exists. Molecular imaging using 89Zr-labeled antibodies may overcome these limitations, enabling the visualization of PD-L1 expression in primary and metastatic tumor lesions and providing information on the in vivo accessibility of the PD-L1 target following intravenous administration. Besides, a baseline FDG-PET scan will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age > 18 years at time of study entry, age > 20 years for Japanese subjects.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy of > 12 weeks
5. Adequate normal organ and marrow function as defined below:

   1. Hemoglobin≥ 9.0 mmol/L
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   3. Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   4. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). (This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician)
   5. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   6. Serum creatinine CL>40 mL/min by MDRD
6. Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
7. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
8. Histological proven recurrent or metastatic squamous cell cancer of the head and neck
9. At least one lesion with a tumor size ≥1 cm

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Previous enrollment in the present study
2. Participation in another clinical study with an investigational product during the last 4 weeks
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
4. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
5. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug 28 days prior to the first dose of study drug for subjects who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C).
6. Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
8. Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)
9. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
10. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
11. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
12. History of primary immunodeficiency
13. History of allogeneic organ transplant
14. History of hypersensitivity to durvalumab or any excipients
15. History of hypersensitivity to the combination or comparator agent (If applicable)
16. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
17. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
18. History of leptomeningeal carcinomatosis
19. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
20. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control: Female patient of child-bearing potential

    * Females of childbearing potential who are sexually active with a non sterilized male partner must use at least 1 highly effective method of contraception (Table 1) from the time of screening and must agree to continue using such precautions for 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy (based on 5x the half-life of durvalumab or tremelimumab). Non-sterilized male partners of a female patient must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Not engaging in sexual activity for the total duration of the drug treatment and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period.
    * Male patients with a female partner of childbearing potential. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from screening through 180 days after receipt of the final dose of durvalumab + tremelimumab combination therapy or 90 days after receipt of the final dose of durvalumab monotherapy. Not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period.
21. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
22. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Tumor uptake of 89Zr-durvalumab | 1 year
  standardized uptake values (SUV) of 89Zr-durvalumab uptake in tumor lesions will be measured.

SECONDARY OUTCOMES:
To assess the potential of PD-L1 PET imaging to predict disease control rate of patients with recurrent or advanced head and neck cancer treated with durvalumab q4w 1500mg iv | 1-2 year
  PD-L1 PET imaging performed with the optimal dose as assessed in part 1 of the study
Correlation between tumor uptake of 89Zr-durvalumab and PD-L1 expression as determined immunohistochemically | 1-2 years
  PD-L1 expression performed by Ventana SP263

CONTACTS AND LOCATIONS:
Overall Officials: carla van Herpen, Prof, Principal Investigator — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - UMC Groningen, Groningen
  - Leiden UMC, Leiden
  - Radboudumc, Nijmegen